CLINICAL TRIAL: NCT02525419
Title: Effects of Intermittent Fasting and Caloric Restriction on Total and Regional Body Composition, Cardiometabolic, Oxidative Stress & Plasma Toxin Biomarkers, and Energy Metabolism in Overweight/Obese Men and Women
Brief Title: Intermittent Fasting, Caloric Restriction and Body Composition in Obese Men and Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Skidmore College (Other)
Collaborators: Isagenix International LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 1307-347
Record Dates: First submitted 2015-08-12; First posted 2015-08-17 (Estimated); Last update posted 2015-08-24 (Estimated); Status verified 2015-08

CONDITIONS: Weight Loss
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Weight Loss Phase (Experimental): 12 week weight loss phase consisting of High Protein - Intermittent Fast-Low Calorie diet in 43 Obese Men and Women
  Interventions: Behavioral: Weight Loss Phase
- Weight Loss Maintenance Phase (Experimental): 52 week weight loss maintenance phase consisting of either High Protein - Intermittent Fast (HP-IF) or Heart Healthy (HH) diet
  Interventions: Behavioral: HP-IF; Behavioral: HH

INTERVENTIONS:
Behavioral: Weight Loss Phase — High Protein, Intermittent Fast, Low Calorie Diet
  Arms: Weight Loss Phase
Behavioral: HP-IF — High Protein, Intermittent Fast
  Arms: Weight Loss Maintenance Phase
Behavioral: HH — Heart Healthy
  Arms: Weight Loss Maintenance Phase

SUMMARY:
This study systematically quantified the effects of intermittent fasting and caloric restriction (IFCR) on total and regional (abdominal) body composition (lean mass and fat mass), blood lipids, toxins, oxidative stress biomarkers, energy expenditure, and substrate utilization in 43 overweight/obese middle-aged men (n=22) and women (n=21). Participants were enrolled in the study as a single cohort and participated in an 12-week trial consisting of two consecutive phases: 1) 1-week baseline, weight maintenance control phase (C), and 2) 11-week weight loss IFCR phase. During the 1 week C phase, volunteers were required to maintain their body weight by consuming their normal food intake; however, during the 11 week IFCR, subjects were instructed to consume 75% of their normal intake to result in a 1-2 lb of body weight loss per week. At the conclusion of the 12 week weight loss study, all 40 participants (3 drop-outs) were invited to enroll in a 12 month follow up study. If they agreed to participate, groups were balanced so there were similar numbers of men and women and were weight-matched. The two groups (n=37, 3 dropped prior to allocation) included: 1) a modified version of the 12 week weight loss intervention that consumes whole foods along with 2 meal replacements (rather than 3) (MR; n=19) or 2) a whole foods diet similar to the Therapeutic Lifestyle Changes diet recommended by the National Institute of Health (TLC, n= 18) and asked to follow these nutritional guidelines ad libitum for the duration of 12 months.

DETAILED DESCRIPTION:
Participants were non-smoking, healthy, but overweight/obese men and women with no known cardiovascular or metabolic diseases as assessed by a medical history and a comprehensive medical examination by their physicians. All participants were sedentary or lightly active (<30 min, 2d/wk of structured physical activity) as assessed by a Physical Activity questionnaire, overweight or obese (BMI>27.5 kg/m2; % body fat>30%), middle aged (30-65 years), and weight stable (+/-2kg) for at least 6 months prior to beginning the study. Individuals with a history of cardiometabolic disease (e.g. diabetes, heart disease, etc) and/or cancer and presently taking medications for these conditions, who are pregnant or may be pregnant, are allergic to milk products or are anorexic or bulimic were excluded from participation. Each participant provided informed written consent in adherence with the Skidmore College Human Subjects review board prior to participation and the study was approved by the Human Subjects Institutional Review Board of Skidmore College. All experimental procedures were performed in accordance with the Federal Wide Assurance and related New York State regulations, which are consistent with the National Commission for the Protection of Human Subjects of Biomedical and Behavioral Research and in agreement with the Helsinki Declaration as revised in 1983.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking, healthy, but overweight/obese men and women with no known cardiovascular or metabolic diseases as assessed by a medical history and a comprehensive medical examination by their physicians
* Sedentary or lightly active (<30 min, 2d/wk of structured physical activity) as assessed by a Physical Activity questionnaire
* Overweight or obese (BMI>27.5 kg/m2; % body fat>30%)
* Weight stable (+/-2kg) for at least 6 months prior to beginning the study

Exclusion Criteria:

* History of cardiometabolic disease (e.g. diabetes, heart disease, etc) and/or cancer and presently taking medications for these conditions
* Pregnant or may be pregnant, are allergic to milk products or are anorexic or bulimic

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2013-08; Primary Completion 2014-11 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Change in Total Body Fat, kg | Baseline, 12 week, 64 weeks
  Quantitative measure of total body fat using the iDXA (dual x-ray absorptiometry)

SECONDARY OUTCOMES:
Change in Serum Toxins | Baseline, 12 weeks, 64 weeks
  Blood Draw
Change in Resting Energy Metabolism | Baseline, 12 weeks, 64 weeks
  indirect Calorimetry
Change in Body Weight, kg | Baseline, 12 week, 64 weeks
  Total body weight measurement

CONTACTS AND LOCATIONS:
Overall Officials: Paul Arciero, Doctorate, Principal Investigator — Faculty
Locations (1):
- Human Nutrition and Metabolism Laboratory, Saratoga Springs, New York, United States

REFERENCES:
- [Derived] Allaf M, Elghazaly H, Mohamed OG, Fareen MFK, Zaman S, Salmasi AM, Tsilidis K, Dehghan A. Intermittent fasting for the prevention of cardiovascular disease. Cochrane Database Syst Rev. 2021 Jan 29;1(1):CD013496. doi: 10.1002/14651858.CD013496.pub2. PMID 33512717